CLINICAL TRIAL: NCT03409887
Title: Effect of Intraorifice Barrier on Healing of Apical Periodontitis: A Randomized Clinical Study
Brief Title: Effect of Intraorifice Barrier on Healing of Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gaurav Kumar
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-01

CONDITIONS: Apical Periodontitis
Keywords: root canal treatment, intraorifice barrier.
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intraorifice Group (Experimental): Intraorifice barrier of GIC.
  Interventions: Procedure: Intraorifice barrier of GIC
- Base Group (Experimental): Base of GIC
  Interventions: Procedure: Base of GIC
- Control Group (Active Comparator): Direct composite restoration
  Interventions: Procedure: Direct composite restoration

INTERVENTIONS:
Procedure: Intraorifice barrier of GIC — After primary root canal treatment, Glass Ionomer Cement (KetacTM Molar, 3M ESPE) applied as intraorifice barrier 3mm inside canal from root canal orifice in first group, as 2mm base on floor of pulp chamber in second group and direct composite restoration in 3rd group without Intraorifice barrier or base.
  Arms: Intraorifice Group
Procedure: Base of GIC — After primary root canal treatment, Glass Ionomer Cement (KetacTM Molar, 3M ESPE) applied as intraorifice barrier 3mm inside canal from root canal orifice in first group, as 2mm base on floor of pulp chamber in second group and direct composite restoration in 3rd group without Intraorifice barrier or base.
  Arms: Base Group
Procedure: Direct composite restoration — After primary root canal treatment, Glass Ionomer Cement (KetacTM Molar, 3M ESPE) applied as intraorifice barrier 3mm inside canal from root canal orifice in first group, as 2mm base on floor of pulp chamber in second group and direct composite restoration in 3rd group without Intraorifice barrier or base.
  Arms: Control Group

SUMMARY:
Based on various in-vitro studies intraorifice barrier has been suggested as an effective mean to provide seal against coronal microleakage. This study intends to clinically investigate efficacy of intraorifice barrier in healing of apical periodontitis.

DETAILED DESCRIPTION:
INTRODUCTION

Coronal leakage is considered significant factor for failure of endodontic treatment. In an array of retrospective studies significant number of cases were reported of apical periodontitis in teeth with unsatisfactory coronal seal as compared to the ones with clinically/radiographically acceptable coronal restoration. Gutta-percha and sealer alone used routinely as root canal obturating material is found to be ineffective to guard against microleakage. Even clinically acceptable root filling allow penetration of bacteria and their products in as less as three days and contribute to eventual treatment failure. This breach of seal in coronal segment of obturated root canal may significantly jeopardize endodontic treatment outcome.

Roghanizad suggested placement of intraorifice barrier to augment coronal seal in endodontically treated teeth. In his study teeth with intraorifice barriers leaked significantly less than the control group where no such barrier was placed. Since then numerous studies have established supremacy of intraorifice barrier and sealing of floor of pulp chamber in preventing coronal microleakage than the one without it. Various materials have been tested as intraorifice barrier. Some studies have reported no difference amongst materials.while other found better performance of MTA over composite and GIC ; GIC over Polycarboxylate cement and Flowable composite.and resilon also composite was found superior over MTA and Cavit and Cavit and IRM.

Various methodology has been employed to study coronal microleakage viz dye penetration ; bacterial penetration ; fluid filtration and glucose molecule penetration.

Intraorifice barrier apart from enhancing probability of success of endodontic treatment may also augment periodontal therapy as intra pulpal infection is known to contribute in worsening of periodontal health by promoting marginal bone loss and pocket formation. Importance of base has also been stressed by Hommez et al who in retrospective study found higher incidence of apical periodontitis in cases where base was absent even though endodontic treatment was adequate.

MATERIALS AND METHODOLOGY:

This study is conducted in the department of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences, Rohtak. Study subjects were obtained from the pool of OPD patients in the Department of Conservative Dentistry and Endodontics, PGIDS, Rohtak.

Prior to treatment a thorough clinical and radiological examination was carried out. A thorough history was taken from each patient. Prior informed consent was taken after explaining the procedure, risk and benefits.

Mature mandibular permanent molar with diagnosis of apical periodontitis (as confirmed clinically & by periapical radiograph) were chosen for the study.

All periapical radiographs were exposed by using constant kVP, mA and exposure time (70 KVP, 8 mA, 0.8 sec.) After initial periodontal therapy, administration of local anesthesia, rubber dam isolation of the involved tooth was done.

Caries excavation was done and access cavity was prepared using carbide burs in high speed handpiece with copious irrigation. Debridement of the pulp chamber was done and all canal orifices were identified. Negotiation of canals was done. Working length was determined using root ZX apex locator and were verified radiographically.

After creating glide path with #15 k-file, Revo-S (Micro Mega, Besancon, France) instruments were used in sequence suggested by manufacturer with a rotational speed of 350 rpm in gentle in-out motion. The torque was adjusted to 2.5 Ncm, and a crown-down approach was selected. Once, the instrument had negotiated to the end of the canal and had rotated freely, it was removed.

Irrigation was carried out using 5 mL of a 5.25% NaOCl solution between files. After preparation, the root canals were irrigated with 5 mL 17% EDTA for 3 minutes to remove smear layer, followed by 5 mL 5.25% NaOCl. The final irrigation was done with 5 mL distilled water.

The root canals were dried using paper points and filled with laterally condensed gutta-percha (Meta Biomed Co Ltd, Korea) and Roth R-801 sealer (Roth International Drug Co., Chicago, Ill) mixed according to manufacturers' instruction

Gutta-percha was cut with a heated instrument and vertically condensed right at the orifice opening of the canals. The teeth were randomly divided into 3 experimental groups as follows :

1. Group I: intraorifice barrier of glass-ionomer cement (KetacTM Molar, 3M ESPE) placed 3mm in the canal from root canal orifice.
2. Group II: base of 2mm of glass-ionomer cement (KetacTM Molar, 3M ESPE) placed on the floor of the pulp chamber.
3. Group III: control group with neither intraorifice barrier placed nor base applied.

In group I: The gutta-percha was removed 3mm from the coronal portion of the canal with hot plugger. Excess root canal sealer was removed with sterilized alcohol-wet cotton pellets. Glass Ionomer Cement was applied inside canal and condensed as well as 2mm thick uniform base on the floor of the pulp chamber.

In group II 2mm thick base of Glass Ionomer Cement was applied uniformly on the floor of the pulp chamber with plastic instrument.

Final composite restoration was placed in all groups according to the manufacturer's instructions. Periodontal therapy in the form of scaling and root planning was done on the day endodontic treatment was completed.

Follow up clinical and radiographic examination was carried out at 3, 6, 9 & 12 month period.

ELIGIBILITY:
Inclusion Criteria:

1. Mature permanent mandibular molars.
2. Pulpal necrosis as confirmed by negative response to pulp sensibility test (cold and electric pulp test) ;
3. Radiographic evidence of apical periodontitis in the form of periapical radiolucency (size not more than 2 × 2mm);

Exclusion Criteria:

1. Younger than 18 years;
2. Pregnant, diabetic, or immunocompromised;
3. Having a positive history of antibiotic use within the past month or require antibiotic premedication for dent treatment (including infective endocarditis or prosthetic joint prophylaxis);
4. Teeth having previous root fillings, unrestorable teeth, fractured/perforated roots, grade 3 mobility, and his of recent periodontal therapy (within previous 6 months);

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-10-14 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical success | Baseline to one year
  Success was defined as absence of signs and symptoms

SECONDARY OUTCOMES:
Radiographic Success | Baseline to one year
  Absence of periapical alterations (radiolucency at furcal or periapical region).

IPD SHARING:
Plan to Share IPD: No